CLINICAL TRIAL: NCT02667587
Title: A Randomized Phase 3 Single Blind Study of Temozolomide Plus Radiation Therapy Combined With Nivolumab or Placebo in Newly Diagnosed Adult Subjects With MGMT-Methylated (Tumor O6-methylguanine DNA Methyltransferase) Glioblastoma
Brief Title: An Investigational Immuno-therapy Study of Temozolomide Plus Radiation Therapy With Nivolumab or Placebo, for Newly Diagnosed Patients With Glioblastoma (GBM, a Malignant Brain Cancer)
Acronym: CheckMate548
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CA209-548; 2015-004722-34 (EudraCT Number)
Expanded Access: NCT02475382 (No longer available)
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Results first posted 2022-02-03 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Brain Neoplasms
MeSH Terms: conditions — Brain Neoplasms | interventions — Nivolumab; Temozolomide; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab + Temozolomide + Radiotherapy (Experimental): Nivolumab: specified dose on specified days; IV (intravenous) infusion Temozolomide: 75 mg (milligram)/meter squared daily during Radiotherapy, 4 week treatment break, 150 mg/meter squared Day 1-5 for Cycle 1 and increased to 200 mg/meter squared Day 1-5 for Cycle2-Cycle 6 as tolerated; orally (additional cycles may be permitted with approval of sponsor) Radiotherapy: 2 gray units (joule of radiation energy per kilogram) 5 times per week for 6 weeks
  Interventions: Drug: Nivolumab; Drug: Temozolomide; Radiation: Radiotherapy
- Nivolumab placebo + Temozolomide + Radiotherapy (Placebo Comparator): Nivolumab Placebo: specified dose on specified days; IV infusion Temozolomide: 75 mg/meter squared daily during Radiotherapy, 4 week treatment break, 150 mg/meter squared Day 1-5 for Cycle 1 and increased to 200 mg/meter squared Day 1-5 for Cycle2-Cycle 6 as tolerated; orally (additional cycles may be permitted with approval of sponsor) Radiotherapy: 2 gray units 5x/week x 6 weeks
  Interventions: Drug: Temozolomide; Radiation: Radiotherapy; Other: Nivolumab Placebo

INTERVENTIONS:
Drug: Nivolumab
  Other Names: Opdivo; Nivo; N; BMS-936558
  Arms: Nivolumab + Temozolomide + Radiotherapy
Drug: Temozolomide
  Other Names: Temodar; TMZ; Temodal; Temcad
Radiation: Radiotherapy
  Other Names: RT
Other: Nivolumab Placebo
  Arms: Nivolumab placebo + Temozolomide + Radiotherapy

SUMMARY:
The purpose of this study is to evaluate patients with glioblastoma that is MGMT-methylated (the MGMT gene is altered by a chemical change). Patients will receive temozolomide plus radiation therapy. They will be compared to patients receiving nivolumab in addition to temozolomide plus radiation therapy.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Males and Females, age ≥ 18 years old
* Newly diagnosed brain cancer or tumor called glioblastoma or GBM
* Karnofsky performance status of ≥ 70 (able to take care of self)
* Substantial recovery from surgery resection
* Tumor test result shows MGMT methylated or indeterminate tumor subtype

Exclusion Criteria:

* Biopsy-only of GBM with less than 20% of tumor removed
* Prior treatment for GBM (other than surgical resection)
* Any known tumor outside of the brain
* Recurrent or secondary GBM
* Active known or suspected autoimmune disease

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2024-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (123):
- United States (35):
  - Local Institution - 0023, Birmingham, Alabama
  - Local Institution - 0003, Phoenix, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Local Institution - 0010, Los Angeles, California
  - Local Institution - 0128, Sacramento, California
  - Local Institution - 0029, San Diego, California
  - Local Institution - 0006, San Francisco, California
  - Local Institution - 0004, New Haven, Connecticut
  - Local Institution - 0031, Washington D.C., District of Columbia
  - Local Institution - 0087, Miami, Florida
  - Local Institution - 0030, Tampa, Florida
  - Local Institution - 0022, Chicago, Illinois
  - Local Institution - 0060, Westwood, Kansas
  - Local Institution - 0018, Louisville, Kentucky
  - Local Institution - 0020, Baltimore, Maryland
  - Local Institution - 0011, Boston, Massachusetts
  - Local Institution - 0028, Boston, Massachusetts
  - Local Institution - 0035, Detroit, Michigan
  - Local Institution - 0002, St Louis, Missouri
  - Local Institution - 0017, Edison, New Jersey
  - Local Institution - 0012, Hackensack, New Jersey
  - Local Institution - 0015, New York, New York
  - Local Institution - 0024, New York, New York
  - Local Institution - 0032, Charlotte, North Carolina
  - Preston Robert Tisch Brain Tumor Center at Duke University, Durham, North Carolina
  - Local Institution - 0001, Cleveland, Ohio
  - Local Institution - 0027, Columbus, Ohio
  - Local Institution - 0098, Allentown, Pennsylvania
  - Local Institution - 0016, Philadelphia, Pennsylvania
  - Local Institution - 0021, Charleston, South Carolina
  - Erlanger Oncology & Hematology - Univ. of TN, Chattanooga, Tennessee
  - Local Institution - 0008, Nashville, Tennessee
  - Local Institution - 0025, Dallas, Texas
  - Local Institution - 0009, Salt Lake City, Utah
  - Local Institution - 0005, Seattle, Washington
- Australia (5):
  - Local Institution - 0049, Liverpool, New South Wales
  - Local Institution - 0052, St Leonards, New South Wales
  - Local Institution - 0050, Heidelberg, Victoria
  - Local Institution - 0051, Prahran, Victoria
  - Local Institution - 0122, Nedlands, Western Australia
- Austria (2):
  - Local Institution - 0062, Linz
  - Local Institution - 0061, Vienna
- Belgium (3):
  - Local Institution - 0070, Brussels
  - Local Institution - 0069, Brussels
  - Local Institution - 0071, Leuven
- Canada (3):
  - Local Institution - 0046, Vancouver, British Columbia
  - Local Institution - 0048, Toronto, Ontario
  - Local Institution - 0047, Montreal, Quebec
- Denmark (2):
  - Local Institution - 0084, Copenhagen
  - Local Institution - 0085, Odense
- France (8):
  - Local Institution - 0043, Lille
  - Local Institution - 0041, Lyon
  - Local Institution - 0040, Marseille
  - Local Institution - 0042, Nancy
  - Local Institution - 0038, Paris
  - Local Institution - 0039, Paris
  - Local Institution - 0044, Rennes
  - Local Institution - 0045, Toulouse
- Germany (11):
  - Local Institution - 0055, Bonn
  - Local Institution - 0131, Cologne
  - Local Institution - 0123, Erlangen
  - Local Institution - 0053, Frankfurt am Main
  - Local Institution - 0124, Freiburg im Breisgau
  - Local Institution - 0057, Hamburg
  - Local Institution - 0056, Heidelberg
  - Local Institution - 0130, Munich
  - Local Institution - 0054, Münster
  - Local Institution - 0058, Regensburg
  - Local Institution - 0059, Tübingen
- Israel (2):
  - Local Institution - 0094, Petah Tikva
  - Local Institution - 0093, Tel Aviv
- Italy (6):
  - Local Institution - 0088, Bologna
  - Local Institution - 0089, Milan
  - Local Institution - 0092, Padua
  - Local Institution - 0127, Rozzano (milano)
  - Local Institution - 0090, Siena
  - Local Institution - 0091, Torino
- Japan (21):
  - Local Institution - 0110, Nagoya, Aichi-ken
  - Local Institution - 0099, Chiba, Chiba
  - Local Institution - 0100, Hiroshima, Hiroshima
  - Local Institution - 0101, Sapporo, Hokkaido
  - Local Institution - 0105, Kobe, Hyōgo
  - Local Institution - 0116, Tsukuba, Ibaraki
  - Local Institution - 0103, Kanazawa, Ishikawa-ken
  - Local Institution - 0102, Kagoshima, Kagoshima-ken
  - Local Institution - 0118, Sagamihara-shi, Kanagawa
  - Local Institution - 0106, Kumamoto, Kumamoto
  - Local Institution - 0120, Okayama, Okayama-ken
  - Local Institution - 0104, Hirakata-shi, Osaka
  - Local Institution - 0112, Suita, Osaka
  - Local Institution - 0121, Hidaka-shi, Saitama
  - Local Institution - 0114, Bunkyo-ku, Tokyo
  - Local Institution - 0111, Chuo-ku, Tokyo
  - Local Institution - 0107, Mitaka-shi, Tokyo
  - Local Institution - 0115, Shinjuku-ku, Tokyo
  - Local Institution - 0117, Yamagata, Yamagata
  - Local Institution - 0109, Kyoto
  - Local Institution - 0108, Kyoto
- Netherlands (4):
  - Local Institution - 0073, Rotterdam, South Holland
  - Local Institution - 0075, Amsterdam
  - Local Institution - 0074, Groningen
  - Local Institution - 0072, Utrecht
- Local Institution - 0083, Oslo, Norway
- Poland (2):
  - Local Institution - 0086, Gdansk
  - Local Institution - 0132, Warsaw
- Russia (2):
  - Local Institution - 0095, Moscow
  - Local Institution - 0097, Moscow
- Spain (7):
  - Local Institution - 0126, Badalona-barcelona
  - Local Institution - 0078, Barcelona
  - Local Institution - 0125, Barcelona
  - Local Institution - 0077, Madrid
  - Local Institution - 0076, Madrid
  - Local Institution - 0080, Santiago Compostela
  - Local Institution - 0079, Valencia
- Sweden (2):
  - Local Institution - 0081, Lund
  - Local Institution - 0082, Solna
- Switzerland (3):
  - Local Institution - 0065, Geneva
  - Local Institution - 0064, Lausanne
  - Local Institution - 0063, Zurich
- United Kingdom (4):
  - Local Institution - 0066, Manchester, Greater Manchester
  - Local Institution - 0119, Sutton, Surrey
  - Local Institution - 0068, Glasgow
  - Local Institution - 0067, London

REFERENCES:
- [Derived] Lim M, Weller M, Idbaih A, Steinbach J, Finocchiaro G, Raval RR, Ansstas G, Baehring J, Taylor JW, Honnorat J, Petrecca K, De Vos F, Wick A, Sumrall A, Sahebjam S, Mellinghoff IK, Kinoshita M, Roberts M, Slepetis R, Warad D, Leung D, Lee M, Reardon DA, Omuro A. Phase III trial of chemoradiotherapy with temozolomide plus nivolumab or placebo for newly diagnosed glioblastoma with methylated MGMT promoter. Neuro Oncol. 2022 Nov 2;24(11):1935-1949. doi: 10.1093/neuonc/noac116. PMID 35511454
- [Derived] Woroniecka K, Fecci PE. Immuno-synergy? Neoantigen vaccines and checkpoint blockade in glioblastoma. Neuro Oncol. 2020 Sep 29;22(9):1233-1234. doi: 10.1093/neuonc/noaa170. No abstract available. PMID 32691060
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 716 participants were randomized into the study, 709 participants received study treatment
Groups:
- Radiotherapy, Temozolomide Plus Nivolumab: Radiotherapy: A total dose of 60 Gy [Gray (radiotherapy dose)], in 2 Gy daily fractions on 5 days/week, will be administered in 6 weeks (30 fractions).
  Nivolumab: 240 mg administered intravenously (IV) as a 30 minute infusion every 2 weeks for 8 doses followed by nivolumab 480 mg as a 30 minute infusion every 4 weeks beginning after 8 doses
  Temozolomide: 75 mg/m2 orally daily during radiation therapy followed by 4 week break then 6 (28-day) cycles temozolomide on Days 1-5 at 150 mg/m2 in Cycle 1 increasing to 200 mg/m2 as tolerated up to 6 cycles.
- Radiotherapy, Temozolomide Plus Placebo: Radiotherapy: A total dose of 60 Gy [Gray (radiotherapy dose)], in 2 Gy daily fractions on 5 days/week, will be administered in 6 weeks (30 fractions).
  Placebo: administered intravenously (IV) as a 30 minute infusion every 2 weeks for 8 doses followed by a 30 minute infusion every 4 weeks beginning after 8 doses
  Temozolomide: 75 mg/m2 orally daily during radiation therapy followed by 4 week break then 6 (28-day) cycles temozolomide on Days 1-5 at 150 mg/m2 in Cycle 1 increasing to 200 mg/m2 as tolerated up to 6 cycles.
Period: Pre-Treatment
Arm/Group | Radiotherapy, Temozolomide Plus Nivolumab | Radiotherapy, Temozolomide Plus Placebo
Started | 358 | 358
Completed | 354 | 355
Not Completed | 4 | 3
Not completed — Not reported | 1 | 0
Not completed — Participant no longer meets study criteria | 2 | 2
Not completed — Participant withdrew consent | 0 | 1
Not completed — Adverse event unrelated to study drug | 1 | 0
Period: End of Treatment
Arm/Group | Radiotherapy, Temozolomide Plus Nivolumab | Radiotherapy, Temozolomide Plus Placebo
Started | 355 (1 participant was randomized to Radiotherapy, Temozolomide plus Placebo but received Radiotherapy, Temozolomide plus Nivolumab.) | 354 (1 participant was randomized to Radiotherapy, Temozolomide plus Placebo but received Radiotherapy, Temozolomide plus Nivolumab.)
Completed | 0 | 0
Not Completed | 355 | 354
Not completed — Disease Progression | 193 | 226
Not completed — Study Drug Toxicity | 75 | 19
Not completed — Death | 2 | 1
Not completed — Adverse Event Unrelated to Study Drug | 19 | 20
Not completed — participant request to discontinue treatment | 33 | 35
Not completed — participant withdrew consent | 5 | 6
Not completed — Lost to Follow-up | 1 | 2
Not completed — maximum clinical benefit | 4 | 4
Not completed — poor or non compliant | 0 | 1
Not completed — participant no longer meets study criteria | 1 | 1
Not completed — administrative reason by sponsor | 1 | 29
Not completed — other reasonse | 21 | 10

BASELINE CHARACTERISTICS:
Population: Demographic characteristics are based off all randomized participants
Groups:
- Radiotherapy, Temozolomide Plus Nivolumab: Nivolumab: specified dose on specified days; IV (intravenous) infusion Temozolomide: 75 mg (milligram)/meter squared daily during Radiotherapy, 4 week treatment break, 150 mg/meter squared Day 1-5 for Cycle 1 and increased to 200 mg/meter squared Day 1-5 for Cycle2-Cycle 6 as tolerated; orally (additional cycles may be permitted with approval of sponsor) Radiotherapy: 2 gray units (joule of radiation energy per kilogram) 5 times per week for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Radiotherapy, Temozolomide Plus Nivolumab | Radiotherapy, Temozolomide Plus Placebo | Total
Number analyzed (Participants) | 358 | 358 | 716
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (12.2) | 58.7 (11.4) | 58.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 161 | 314
  Male | 205 | 197 | 402
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 11 | 18
  Not Hispanic or Latino | 171 | 178 | 349
  Unknown or Not Reported | 180 | 169 | 349
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 301 | 318 | 619
  Black or African American | 4 | 4 | 8
  Asian | 35 | 33 | 68
  Other | 17 | 3 | 20
  Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Determined by BICR
Description: The time from randomization to the date of the first documented tumor progression or death by any cause. PFS will be determined by a Blinded Independent Central Review (BICR) assessed based on Radiologic Assessment in Neuro-Oncology (RANO) criteria. Specifically, RANO response criteria indicates that within the first 12 weeks of completion of radiotherapy, progression can only be assessed if the majority of the new enhancement is outside of the radiation field or if there is pathologic confirmation of progressive disease.
Time Frame: From randomization to the date of the first documented tumor progression or death by any cause. (up to approximately 4.5 years)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radiotherapy, Temozolomide Plus Nivolumab | Radiotherapy, Temozolomide Plus Placebo
Number analyzed (Participants) | 358 | 358
Months | 10.64 [8.90 to 11.79] | 10.32 [9.69 to 12.45]
Statistical Analysis 1: Comparison: Radiotherapy, Temozolomide Plus Nivolumab; Test type: Superiority; Cox Proportional Hazard = 1.06, 95% CI 2-sided [0.90 to 1.25]

2. Primary Outcome: Overall Survival (OS)
Description: The time from the date of randomization to the date of death. who have not died by the end of the study will be censored to last known date alive. OS is assessed in the randomized population with no corticosteroids at baseline population and in the overall randomized population.
Time Frame: From randomization to date of death (up to approximately 4.5 years)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radiotherapy, Temozolomide Plus Nivolumab | Radiotherapy, Temozolomide Plus Placebo
Number analyzed (Participants) | 358 | 358
Months
  All randomized participants | 28.91 [24.38 to 31.57] | 32.07 [29.37 to 33.77]
  All randomized participants without baseline corticosteroids: number analyzed (Participants) | 246 | 262
  All randomized participants without baseline corticosteroids | 31.34 [28.62 to 34.76] | 32.99 [31.01 to 35.09]
Statistical Analysis 1: Comparison: Radiotherapy, Temozolomide Plus Nivolumab; All Randomized No Baseline Corticosteroids Participants; Test type: Superiority; p = 0.3402, Log Rank; Cox Proportional Hazard = 1.12, 96.39% CI 2-sided [0.87 to 1.43]
Statistical Analysis 2: Comparison: Radiotherapy, Temozolomide Plus Nivolumab; All Randomized Participants; Test type: Superiority; Cox Proportional Hazard = 1.10, 95% CI 2-sided [0.91 to 1.33]

3. Secondary Outcome: Overall Survival (OS) Rates at 12 Months
Description: Overall Survival (OS) rate is defined as the percentage of participants surviving at 12 months
Time Frame: From randomization to 12 months after first dose
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy, Temozolomide Plus Nivolumab | Radiotherapy, Temozolomide Plus Placebo
Number analyzed (Participants) | 358 | 358
percentage of participants | 82.7 [78.3 to 86.3] | 87.7 [83.8 to 90.8]

4. Secondary Outcome: Overall Survival (OS) Rates at 24 Months
Description: Overall Survival (OS) rate is defined as the percentage of participants surviving at 24 months
Time Frame: From randomization to 24 months after first dose
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy, Temozolomide Plus Nivolumab | Radiotherapy, Temozolomide Plus Placebo
Number analyzed (Participants) | 358 | 358
percentage of participants | 55.9 [50.5 to 61.0] | 63.3 [58 to 68.2]

5. Secondary Outcome: Progression Free Survival (PFS) Based on Investigator Assessment
Description: The time from randomization to the date of the first documented tumor progression or death by any cause. PFS will be determined by investigator assessment based Radiologic Assessment in Neuro-Oncology (RANO) criteria. Specifically, RANO response criteria indicates that within the first 12 weeks of completion of radiotherapy, progression can only be assessed if the majority of the new enhancement is outside of the radiation field or if there is pathologic confirmation of progressive disease.
Time Frame: as for outcome 1
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radiotherapy, Temozolomide Plus Nivolumab | Radiotherapy, Temozolomide Plus Placebo
Number analyzed (Participants) | 358 | 358
Months | 14.09 [12.62 to 16.56] | 15.18 [13.11 to 17.12]

6. Post Hoc Outcome: Progression-free Survival (PFS) Determined by BICR - Extended Collection
Description: as for outcome 1
Time Frame: From randomization to the date of the first documented tumor progression or death by any cause. (up to approximately 82 Months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radiotherapy, Temozolomide Plus Nivolumab | Radiotherapy, Temozolomide Plus Placebo
Number analyzed (Participants) | 358 | 358
Months | 9.89 [8.31 to 11.60] | 10.25 [9.46 to 12.09]
Statistical Analysis 1: Comparison: Radiotherapy, Temozolomide Plus Nivolumab; Test type: Superiority; Cox Proportional Hazard = 1.18, 95% CI 2-sided [0.99 to 1.40]

7. Post Hoc Outcome: Overall Survival (OS) - Extended Collection
Description: The time from the date of randomization to the date of death. who have not died by the end of the study will be censored to last known date alive. OS is assessed in the randomized population with no corticosteroids at baseline population.
Time Frame: From randomization to date of death (up to approximately 82 Months)
Population: All randomized participants with no baseline corticosteroids
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radiotherapy, Temozolomide Plus Nivolumab | Radiotherapy, Temozolomide Plus Placebo
Number analyzed (Participants) | 246 | 262
Months | 28.94 [24.57 to 31.64] | 31.84 [28.94 to 33.77]
Statistical Analysis 1: Comparison: Radiotherapy, Temozolomide Plus Nivolumab vs Radiotherapy, Temozolomide Plus Placebo; Test type: Superiority; Log Rank; Cox Proportional Hazard = 1.06, 95% CI 2-sided [0.89 to 1.26]

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: (From first dose to last dose + 100 days): Approximately 48 Months All-Cause mortality (From randomization to end of study): Approximately up to 52 months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Radiotherapy, Temozolomide Plus Nivolumab | Radiotherapy, Temozolomide Plus Placebo
All-Cause Mortality (participants affected / at risk) | 263/358 | 255/358
Serious Adverse Events (participants affected / at risk) | 259/355 | 217/354
Other Adverse Events (participants affected / at risk) | 351/355 | 343/354
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy, Temozolomide Plus Nivolumab (N=355) | Radiotherapy, Temozolomide Plus Placebo (N=354)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 1
Pancytopenia (Blood and lymphatic system disorders) | 8 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 7
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 2 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Branchial cyst (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 2
Diabetes insipidus (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 3 | 0
Cataract (Eye disorders) | 1 | 1
Diplopia (Eye disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 1
Iridocyclitis (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Autoimmune colitis (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 5 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 3 | 3
Cyst (General disorders) | 1 | 0
Death (General disorders) | 4 | 3
Drowning (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Gait disturbance (General disorders) | 1 | 1
Gait inability (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 8 | 4
Hyperthermia (General disorders) | 1 | 0
Influenza like illness (General disorders) | 2 | 0
Localised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 16 | 4
Sudden death (General disorders) | 2 | 3
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 3 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1
Haemorrhagic hepatic cyst (Hepatobiliary disorders) | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 3 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 3 | 1
Immunodeficiency (Immune system disorders) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2
Bacterial infection (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 1 | 2
Gastrointestinal infection (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 5 | 1
Influenza (Infections and infestations) | 0 | 2
Intervertebral discitis (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 1
Meningitis aseptic (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 14 | 5
Pneumonia aspiration (Infections and infestations) | 4 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 2
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyometra (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 4 | 1
Septic shock (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 7 | 4
Urosepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 3 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Incision site swelling (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 2
Alanine aminotransferase increased (Investigations) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Influenza A virus test positive (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 6 | 3
White blood cell count decreased (Investigations) | 4 | 1
Adult failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Autoimmune myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Eosinophilic fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 12
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 75 | 73
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 11
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 7
Tumour pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute disseminated encephalomyelitis (Nervous system disorders) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 3 | 5
Brain oedema (Nervous system disorders) | 8 | 7
Central nervous system lesion (Nervous system disorders) | 0 | 1
Central nervous system necrosis (Nervous system disorders) | 0 | 1
Cerebral cyst (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 3
Cerebral ischaemia (Nervous system disorders) | 2 | 3
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 3 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 2
Change in seizure presentation (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 2 | 6
Coma (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 4
Drooling (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 4 | 5
Epilepsy (Nervous system disorders) | 15 | 12
Generalised tonic-clonic seizure (Nervous system disorders) | 2 | 1
Haemorrhage intracranial (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 8 | 6
Hemiparesis (Nervous system disorders) | 7 | 9
Hemiplegia (Nervous system disorders) | 3 | 0
Hydrocephalus (Nervous system disorders) | 10 | 9
Intracranial pressure increased (Nervous system disorders) | 1 | 3
Ischaemic stroke (Nervous system disorders) | 2 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 2
Neurological decompensation (Nervous system disorders) | 0 | 2
Neurological symptom (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Optic neuritis (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 2 | 1
Psychomotor skills impaired (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 48 | 40
Simple partial seizures (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1
Status epilepticus (Nervous system disorders) | 1 | 1
Subdural hygroma (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 2 | 1
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 2
Device malfunction (Product Issues) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 2 | 2
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 5 | 0
Mood altered (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 2
Bladder stenosis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephritis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 13
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Assisted suicide (Surgical and medical procedures) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Euthanasia (Surgical and medical procedures) | 1 | 0
Axillary vein thrombosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 2
Embolism (Vascular disorders) | 5 | 5
Hypotension (Vascular disorders) | 2 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy, Temozolomide Plus Nivolumab (N=355) | Radiotherapy, Temozolomide Plus Placebo (N=354)
Anaemia (Blood and lymphatic system disorders) | 42 | 26
Leukopenia (Blood and lymphatic system disorders) | 20 | 30
Lymphopenia (Blood and lymphatic system disorders) | 43 | 39
Neutropenia (Blood and lymphatic system disorders) | 33 | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 69 | 67
Hypothyroidism (Endocrine disorders) | 28 | 9
Dry eye (Eye disorders) | 18 | 15
Vision blurred (Eye disorders) | 30 | 23
Abdominal pain (Gastrointestinal disorders) | 32 | 27
Constipation (Gastrointestinal disorders) | 163 | 145
Diarrhoea (Gastrointestinal disorders) | 77 | 72
Nausea (Gastrointestinal disorders) | 187 | 159
Stomatitis (Gastrointestinal disorders) | 25 | 9
Vomiting (Gastrointestinal disorders) | 90 | 75
Asthenia (General disorders) | 42 | 40
Chills (General disorders) | 25 | 13
Fatigue (General disorders) | 186 | 176
Gait disturbance (General disorders) | 29 | 34
Malaise (General disorders) | 17 | 18
Oedema peripheral (General disorders) | 30 | 28
Pain (General disorders) | 18 | 9
Pyrexia (General disorders) | 70 | 31
Conjunctivitis (Infections and infestations) | 20 | 12
Nasopharyngitis (Infections and infestations) | 37 | 31
Oral candidiasis (Infections and infestations) | 20 | 12
Upper respiratory tract infection (Infections and infestations) | 21 | 19
Urinary tract infection (Infections and infestations) | 45 | 34
Fall (Injury, poisoning and procedural complications) | 37 | 46
Radiation skin injury (Injury, poisoning and procedural complications) | 35 | 38
Alanine aminotransferase increased (Investigations) | 63 | 39
Aspartate aminotransferase increased (Investigations) | 46 | 16
Blood creatinine increased (Investigations) | 23 | 14
Lymphocyte count decreased (Investigations) | 67 | 62
Neutrophil count decreased (Investigations) | 34 | 40
Platelet count decreased (Investigations) | 75 | 75
Weight decreased (Investigations) | 50 | 33
Weight increased (Investigations) | 13 | 21
White blood cell count decreased (Investigations) | 40 | 44
Decreased appetite (Metabolism and nutrition disorders) | 97 | 87
Hyperglycaemia (Metabolism and nutrition disorders) | 25 | 34
Hypokalaemia (Metabolism and nutrition disorders) | 34 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 61 | 53
Back pain (Musculoskeletal and connective tissue disorders) | 41 | 34
Muscular weakness (Musculoskeletal and connective tissue disorders) | 35 | 28
Myalgia (Musculoskeletal and connective tissue disorders) | 30 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 | 16
Aphasia (Nervous system disorders) | 30 | 32
Cognitive disorder (Nervous system disorders) | 19 | 19
Dizziness (Nervous system disorders) | 47 | 53
Dysgeusia (Nervous system disorders) | 36 | 27
Headache (Nervous system disorders) | 142 | 135
Hemiparesis (Nervous system disorders) | 23 | 25
Memory impairment (Nervous system disorders) | 26 | 36
Paraesthesia (Nervous system disorders) | 26 | 23
Seizure (Nervous system disorders) | 63 | 76
Tremor (Nervous system disorders) | 22 | 26
Anxiety (Psychiatric disorders) | 32 | 34
Confusional state (Psychiatric disorders) | 20 | 21
Depression (Psychiatric disorders) | 30 | 34
Insomnia (Psychiatric disorders) | 54 | 47
Pollakiuria (Renal and urinary disorders) | 18 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 59 | 51
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 | 20
Alopecia (Skin and subcutaneous tissue disorders) | 115 | 109
Dry skin (Skin and subcutaneous tissue disorders) | 24 | 27
Erythema (Skin and subcutaneous tissue disorders) | 29 | 22
Pruritus (Skin and subcutaneous tissue disorders) | 86 | 77
Rash (Skin and subcutaneous tissue disorders) | 85 | 58
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 32 | 13
Hypertension (Vascular disorders) | 29 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT02667587/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT02667587/SAP_001.pdf